CLINICAL TRIAL: NCT01412424
Title: Efficacy and Safety of Oral Octreolin™ in Patients With Acromegaly Who Are Currently Receiving Parenteral Somatostatin Analogs
Brief Title: Efficacy and Safety of Octreotide (MYCAPSSA™ [Formerly Octreolin™]) for Acromegaly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiasma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-ACM-01
Record Dates: First submitted 2011-08-05; First posted 2011-08-09 (Estimated); Results first posted 2015-12-01 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-07

CONDITIONS: Acromegaly
Keywords: acromegaly; IGF-1; growth hormone; Octreolin; octreotide; somatostatin analog
MeSH Terms: conditions — Acromegaly | interventions — Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Octreotide capsules (Experimental): Participants received octreotide capsules orally twice a day for up to 13 months. Dosing started at 40 mg per day (20 in the morning + 20 in the evening) and increased to 60 mg per day (40 in the morning + 20 in the evening) or 80 mg per day (40 in the morning + 40 in the evening) if there was inadequate IGF-1 suppression.
  Interventions: Drug: Octreotide capsules

INTERVENTIONS:
Drug: Octreotide capsules — Octreotide was provided in hard gelatin capsules.
  Other Names: MYCAPSSA™; Formerly known as Octreolin™

SUMMARY:
MYCAPSSA™ (formerly Octreolin™) is a proprietary oral form of the approved injectable medical product octreotide used to treat acromegaly. This study will evaluate the efficacy and safety of MYCAPSSA™ treatment in patients with acromegaly.

DETAILED DESCRIPTION:
The study consisted of 2 periods, a Core Treatment Period of up to 7 months and an optional Extension Treatment Period of up to 6 months, for a total study duration of up to 13 months. The Core Treatment Period consisted of 2 phases, a Dose Escalation Phase of at least 2 months to identify the therapeutic dose for each study participant and a Fixed Dose Phase of 2 to 5 months during which the therapeutic dose was maintained.

Participants were eligible to enter the Fixed Dose Phase of the Core Treatment Period if they were clinically and biochemically controlled. The same criteria were used to allow entry into the voluntary 6-month Extension Treatment Period.

The Core Treatment Period of the study was completed if the participant had at least 2 months of treatment in the Fixed Dose Phase and a total treatment duration of at least 7 months. Participants who elected to continue into the Extension Treatment Period maintained their therapeutic dose during this period. At the end of the study (after the last dose of MYCAPSSA in either the Core Treatment Period or the Extension Treatment Period), there was a 2-week follow-up period for safety assessments.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects, aged 18 to 75 years old, inclusive.
* Subjects with acromegaly defined as documented evidence of growth hormone-secreting pituitary tumor that is abnormally responsive to glucose, or documented elevated insulin-like growth factor-1 (IGF-1), who are currently receiving a stable dose of a somatostatin analog for at least the previous 3 months.
* A serum IGF-1 level < 1.3 x the upper limit of normal (ULN) and a serum growth hormone (GH) level < 2.5 ng/mL.
* Subjects able and willing to comply with the requirements of the protocol.
* Subjects able to swallow capsules.
* Subjects able to understand and sign written informed consent to participate in the study.

Exclusion Criteria:

* Receiving regular injections of a somatostatin analog less frequently than once a month, ie, longer than every 4 weeks.
* Symptomatic cholelithiasis.
* Received pituitary radiotherapy within ten years prior to screening.
* Undergone pituitary surgery within the prior 6 months.
* Any condition that may jeopardize study participation.
* Clinically significant gastrointestinal (GI), renal, or hepatic disease as determined by the Investigator.
* Conditions (eg, bariatric surgery) significantly affecting gastric acidity or emptying.
* Current use (within 1 month) of proton pump inhibitors (PPIs) and current chronic use of H2-antagonists.
* Female patients who are pregnant or lactating.
* Current or recent (< 3 months) therapy with pegvisomant.
* Current or recent (< 2 months) therapy with cabergoline.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2012-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shlomo Melmed, MD, Study Chair — Cedars-Sinai Medical Center
Locations (36):
- Cedars-Sinai Medical Center, Los Angeles, California, United States
- Germany (5):
  - Campus Charité Mitte, Berlin
  - ENDOC Center for Endocrine Tumors, Hamburg
  - Medizinische Klinik Innenstadt, Munich
  - Max Planck Institute of Psychiatry, Munich
  - Praxis for Endocrimology and Diabetology in Oldenburg, Oldenburg
- Hungary (4):
  - Military Hospital, State Health Center 2nd Department of Internal Medicine, Budapest
  - Semmelweiss University, Budapest
  - University of Pecs, Pécs
  - University of Szeged, Szeged
- Italy (3):
  - Servizio di Endocrinologia A.O. Spedali Civili di Brescia, Brescia
  - Dipartimento Clinico Sperimentale di Medicina e Farmacologia, Messina
  - Ospedale Molinette, Torino
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kauno Klinikos, Kaunas
  - Vilnius University Hospital Santariskiu Clinics Center of Endocrinology, Vilnius
- Mexico (3):
  - Unidad de Investigacion Clinica Cardiometabolica de Occidente, Guadalajara Jalisco
  - Instituto Nacional de Neurologia y Neurocirugía - National Institute of Neurology and Neurosurgery, Mexico City
  - Centro Medico ABC, Mexico City
- Netherlands (2):
  - Leiden University Medical Centre, Leiden
  - Erasmus University Medical Center, Rotterdam
- Poland (5):
  - Autonomous Public Clinical Hospital No. 5, Katowice
  - Department of Endocrinology - Jagiellonian University, Krakow, Krakow
  - Clinical Hospital of Medical University in Poznan, Poznan
  - Bielanski Hospital, Warsaw
  - Wroclaw Medical University, Wroclaw
- Romania (2):
  - Endocrinology Institute C.I.Parhon, Bucharest
  - County Emergency Hospital, Sf. Spiridon, Department of Endocrinology, Iași
- Serbia (2):
  - Clinic for Endocrinology, Diabetes and Metabolism Diseases, Clinical Center of Serbia, Belgrade
  - Clinical Center of Vojvodina, Novi Sad
- Slovakia (2):
  - University Hospital Bratislava, Hospital of L.Derer, Bratislava
  - National Institute of Endocrinology and Diabetology, Ľubochňa
- Department of Endocrinology and Diabetes, University Medical Centre, Ljubliana, Slovenia
- United Kingdom (4):
  - University of Warwick - Medical School, Coventry
  - St Bartholomew's Hospital West, London
  - The Christie Hospital NHS Trust, Manchester
  - Oxford Centre for Diabetes, Endocrinology and Metabolism, Oxford

REFERENCES:
- [Derived] Labadzhyan A, Nachtigall LB, Fleseriu M, Gordon MB, Molitch M, Kennedy L, Samson SL, Greenman Y, Biermasz N, Bolanowski M, Haviv A, Ludlam W, Patou G, Strasburger CJ. Oral octreotide capsules for the treatment of acromegaly: comparison of 2 phase 3 trial results. Pituitary. 2021 Dec;24(6):943-953. doi: 10.1007/s11102-021-01163-2. Epub 2021 Jun 25. PMID 34173129
- [Derived] Melmed S, Popovic V, Bidlingmaier M, Mercado M, van der Lely AJ, Biermasz N, Bolanowski M, Coculescu M, Schopohl J, Racz K, Glaser B, Goth M, Greenman Y, Trainer P, Mezosi E, Shimon I, Giustina A, Korbonits M, Bronstein MD, Kleinberg D, Teichman S, Gliko-Kabir I, Mamluk R, Haviv A, Strasburger C. Safety and efficacy of oral octreotide in acromegaly: results of a multicenter phase III trial. J Clin Endocrinol Metab. 2015 Apr;100(4):1699-708. doi: 10.1210/jc.2014-4113. Epub 2015 Feb 9. PMID 25664604
- See also: Sponsor website — http://www.chiasmapharma.com

RESULTS

PARTICIPANT FLOW:
Period: Core Treatment Period
Arm/Group | Octreotide Capsules
Started | 155
Completed | 102
Not Completed | 53
Not completed — Treatment Failure | 24
Not completed — Adverse Event | 21
Not completed — Patient Request | 5
Not completed — Lost to Follow-up | 2
Not completed — Sponsor Request | 1
Period: Extension Treatment Period
Arm/Group | Octreotide Capsules
Started | 88 (86% of participants who completed the core period voluntarily entered the optional extension period.)
Completed | 82
Not Completed | 6
Not completed — Adverse Event | 2
Not completed — Treatment Failure | 2
Not completed — Patient Request | 2

BASELINE CHARACTERISTICS:
Population: Safety population: All participants enrolled in the study who received any amount of the study drug.
Arm/Group | Octreotide Capsules
Number analyzed (Participants) | 155
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.2 (11.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88
  Male | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 135
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 137
  More than one race | 0
  Unknown or Not Reported | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders at the End of the Core Treatment Period
Description: A responder was defined as a participant with a serum insulin-like growth factor-1 (IGF-1) concentration < 1.3 times the upper limit of normal (adjusted for age and gender) and a growth hormone (GH) concentration < 2.5 ng/mL. The growth hormone concentration was the mean of 5 fasted GH serum concentrations collected at 30 minute intervals for 2 hours, 2 to 4 hours post-octreotide dose. IGF-1 concentration was determined in serum samples taken at the same visits GH concentration was assessed.
Time Frame: End of the core treatment period (up to 7 months)
Population: Modified intent-to-treat population: All enrolled participants who received any amount of study drug and who had at least 1 IGF-1 or GH assessment after the first dose of octreotide.
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Groups:
- Octreotide 40 mg: Participants received octreotide 20 mg orally twice a day for up to 13 months.
- Octreotide 60 mg: Participants received octreotide 40 mg in the morning and octreotide 20 mg in the evening orally for up to 13 months.
- Octreotide 80 mg: Participants received octreotide 40 mg in the morning and octreotide 40 mg in the evening orally for up to 13 months.
- Octreotide 40, 60, or 80 mg - All Participants: Participants received octreotide 40, 60, or 80 mg orally for up to 13 months.
Arm/Group | Octreotide 40 mg | Octreotide 60 mg | Octreotide 80 mg | Octreotide 40, 60, or 80 mg - All Participants
Number analyzed (Participants) | 61 | 33 | 57 | 151
Percentage of responders | 86.9 [83.0 to 98.1] | 66.7 [48.2 to 82.0] | 40.4 [27.6 to 54.2] | 64.9 [58.4 to 74.2]

2. Primary Outcome: Percentage of Responders at the End of the Extension Treatment Period
Description: as for outcome 1
Time Frame: End of the extension treatment period (up to 13 months)
Population: Extension intent-to-treat population: All participants who entered the extension treatment period and received any amount of study drug during the extension treatment period.
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | Octreotide Capsules
Number analyzed (Participants) | 88
Percentage of responders | 78.4 [68.4 to 86.5]

3. Secondary Outcome: Percentage of Participants With Specified IGF-1 and GH Concentrations at Baseline and at the End of the Core Treatment Period
Description: Percentage of participants with the following serum insulin-like growth factor-1 (IGF-1) and growth hormone (GH) concentrations at Baseline and at the end of the core treatment period (ECTP): IGF-1 < 1.3 times the upper limit of normal (ULN) and GH < 5.0 ng/mL, IGF-1 < 1.3 times ULN and GH < 1.0 ng/mL, IGF-1 ≤ 1.0 times ULN and GH < 5.0 ng/mL, IGF-1 ≤ 1.0 times ULN and GH < 2.5 ng/mL, IGF-1 ≤ 1.0 times ULN and GH < 1.0 ng/mL, IGF-1 < 1.3 times ULN, IGF-1 ≤ 1.0 times ULN, GH < 5.0 ng/mL, GH < 2.5 ng/mL, GH < 1.0 ng/mL, IGF-1 ≥ 1.3 times ULN and GH < 2.5 ng/mL, IGF-1 < 1.3 times ULN and GH ≥ 2.5 ng/mL, and IGF-1 ≥ 1.3 times ULN and GH ≥ 2.5 ng/mL. The growth hormone concentration was the mean of 5 fasted GH serum concentrations collected at 30 minute intervals for 2 hours, 2 to 4 hours post-octreotide dose. IGF-1 concentration was determined in serum samples taken at the same visits GH concentration was assessed.
Time Frame: Baseline and the end of the core treatment period (up to 7 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Octreotide Capsules
Number analyzed (Participants) | 151
Percentage of participants
  IGF-1 < 1.3 & GH < 5.0: Baseline | 91.4
  IGF-1 < 1.3 & GH < 5.0: ECTP | 65.6
  IGF-1 < 1.3 & GH < 1.0: Baseline | 62.9
  IGF-1 < 1.3 & GH < 1.0: ECTP | 53.0
  IGF-1 ≤ 1.0 & GH < 5.0: Baseline | 63.6
  IGF-1 ≤ 1.0 & GH < 5.0: ECTP | 35.8
  IGF-1 ≤ 1.0 & GH < 2.5: Baseline | 61.6
  IGF-1 ≤ 1.0 & GH < 2.5: ECTP | 35.8
  IGF-1 ≤ 1.0 & GH < 1.0: Baseline | 43.0
  IGF-1 ≤ 1.0 & GH < 1.0: ECTP | 31.8
  IGF-1 < 1.3: Baseline | 91.4
  IGF-1 < 1.3: ECTP | 66.9
  IGF-1 ≤ 1.0: Baseline | 63.6
  IGF-1 ≤ 1.0: ECTP | 37.1
  GH < 5.0: Baseline | 100.0
  GH < 5.0: ECTP | 97.4
  GH < 2.5: Baseline | 96.0
  GH < 2.5: ECTP | 94.7
  GH < 1.0: Baseline | 66.2
  GH < 1.0: ECTP | 77.5
  IGF-1 ≥ 1.3 & GH < 2.5: Baseline | 7.3
  IGF-1 ≥ 1.3 & GH < 2.5: ECTP | 29.8
  IGF-1 < 1.3 & GH ≥ 2.5: Baseline | 2.6
  IGF-1 < 1.3 & GH ≥ 2.5: ECTP | 0.7
  IGF-1 ≥ 1.3 & GH ≥ 2.5: Baseline | 1.3
  IGF-1 ≥ 1.3 & GH ≥ 2.5: ECTP | 2.0

4. Secondary Outcome: Maintenance of Response During the Fixed Dose Phase of the Core Treatment Period
Description: Maintenance of response during the fixed dose phase of the core treatment period was defined as the percentage of participants with an insulin-like growth factor-1 (IGF-1) concentration < 1.3 times the upper limit of normal at the beginning of the fixed dose phase of the core treatment period and at the end of the core treatment period. IGF-1 concentration was determined in serum samples taken at the same visits growth hormone concentration was assessed.
Time Frame: Beginning of the fixed dose phase of the core treatment period and the end of the core treatment period (up to 7 months)
Population: Fixed dose population: All enrolled participants who received any amount of study drug, who had at least 1 IGF-1 or GH assessment after the first dose of octreotide, and who entered the fixed dose phase of the core treatment period.
Measure: Number; unit: Percentage of participants
Arm/Group | Octreotide Capsules
Number analyzed (Participants) | 110
Percentage of participants
  Beginning of the FDP of the CTP | 82.7
  End of the CTP | 80.0

5. Secondary Outcome: Percentage of Participants With Specified IGF-1 and GH Concentrations at the Beginning and at the End of the Extension Treatment Period
Description: Percentage of participants with the following serum insulin-like growth factor-1 (IGF-1) and growth hormone (GH) concentrations at the beginning (BETP) and at the end (EETP) of the extension treatment period: IGF-1 < 1.3 times the upper level of normal (ULN) and GH < 5.0 ng/mL, IGF-1 < 1.3 times ULN and GH < 1.0 ng/mL, IGF-1 ≤ 1.0 times ULN and GH < 5.0 ng/mL, IGF-1 ≤ 1.0 times ULN and GH < 2.5 ng/mL, IGF-1 ≤ 1.0 times ULN and GH < 1.0 ng/mL, IGF-1 < 1.3 times ULN, IGF-1 ≤ 1.0 times ULN, GH < 5.0 ng/mL, GH < 2.5 ng/mL, GH < 1.0 ng/mL, IGF-1 ≥ 1.3 times ULN and GH < 2.5 ng/mL, IGF-1 < 1.3 times ULN and GH ≥ 2.5 ng/mL, and IGF-1 ≥ 1.3 times ULN and GH ≥ 2.5 ng/mL. The growth hormone concentration was the mean of 5 fasted GH serum concentrations collected at 30 minute intervals for 2 hours, 2 to 4 hours post-octreotide dose. IGF-1 concentration was determined in serum samples taken at the same visits GH concentration was assessed.
Time Frame: Beginning and the end of the extension treatment period (up to 6 months)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Octreotide Capsules
Number analyzed (Participants) | 88
Percentage of participants
  IGF-1 < 1.3 & GH < 5.0: BETP | 84.1
  IGF-1 < 1.3 & GH < 5.0: EETP | 79.5
  IGF-1 < 1.3 & GH < 1.0: BETP | 69.3
  IGF-1 < 1.3 & GH < 1.0: EETP | 68.2
  IGF-1 ≤ 1.0 & GH < 5.0: BETP | 48.9
  IGF-1 ≤ 1.0 & GH < 5.0: EETP | 50.0
  IGF-1 ≤ 1.0 & GH < 2.5: BETP | 48.9
  IGF-1 ≤ 1.0 & GH < 2.5: EETP | 50.0
  IGF-1 ≤ 1.0 & GH < 1.0: BETP | 42.0
  IGF-1 ≤ 1.0 & GH < 1.0: EETP | 44.3
  IGF-1 < 1.3: BETP | 84.1
  IGF-1 < 1.3: EETP | 79.5
  IGF-1 ≤ 1.0: BETP | 48.9
  IGF-1 ≤ 1.0: EETP | 50.0
  GH < 5.0: BETP | 100.0
  GH < 5.0: EETP | 97.7
  GH < 2.5: BETP | 98.9
  GH < 2.5: EETP | 95.5
  GH < 1.0: BETP | 83.0
  GH < 1.0: EETP | 83.0
  IGF-1 ≥ 1.3 & GH < 2.5: BETP | 14.8
  IGF-1 ≥ 1.3 & GH < 2.5: EETP | 17.0
  IGF-1 < 1.3 & GH ≥ 2.5: BETP | 0.0
  IGF-1 < 1.3 & GH ≥ 2.5: EETP | 1.1
  IGF-1 ≥ 1.3 & GH ≥ 2.5: BETP | 1.1
  IGF-1 ≥ 1.3 & GH ≥ 2.5: EETP | 3.4

6. Secondary Outcome: Maintenance of Response During the Extension Treatment Period
Description: Maintenance of an insulin-like growth factor-1 (IGF-1) response during the extension treatment period was defined as the percentage of participants with an IGF-1 concentration < 1.3 times the upper limit of normal at the beginning of the extension treatment period and at the end of the extension treatment period. IGF-1 concentration was determined in serum samples taken at the same visits growth hormone concentration was assessed.
Time Frame: Beginning of the extension treatment period and the end of the extension treatment period (up to 13 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Octreotide Capsules
Number analyzed (Participants) | 74
Percentage of participants | 87.8 [78.2 to 94.3]

7. Secondary Outcome: Percentage of Participants With Improved or Maintained Acromegaly Symptoms at the End of the Extension Treatment Period
Description: The severity (absent, mild, moderate, severe) of the 5 acromegaly symptoms headache, perspiration, asthenia, swelling of extremities, and joint pain was assessed at Baseline and at the end of the extension treatment period. The percentage of participants with improved or maintained (no change) acromegaly symptoms from Baseline at the end of the extension treatment period is reported.
Time Frame: Baseline and the end of the extension treatment period (up to 13 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Octreotide Capsules
Number analyzed (Participants) | 88
Percentage of participants
  Maintained | 27 [18.3 to 37.8]
  Improved | 57 [45.8 to 67.3]

8. Secondary Outcome: Percentage of Participants With ≥ 1, 2, or 3 Acromegaly Symptoms at Baseline and at the End of the Extension Treatment Period
Description: Reported is the percentage of participants who had ≥ 1, 2, or 3 of the 5 symptoms of acromegaly (headaches, perspiration, asthenia, swelling of extremities, or joint pain) of any severity (mild, moderate, or severe). This was a post hoc analysis.
Time Frame: Baseline and the end of the extension treatment period (up to 13 months)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Octreotide Capsules
Number analyzed (Participants) | 88
Percentage of participants
  1 Symptom - Baseline | 78
  1 Symptom - End of the extension treatment period | 65
  2 Symptoms - Baseline | 61
  2 Symptoms - End of the extension treatment period | 43
  3 Symptoms - Baseline | 43
  3 Symptoms - End of the extension treatment period | 25

ADVERSE EVENTS:
Description: Safety population: All participants enrolled in the study who received any amount of the study drug.
  The total number of participants with adverse events is greater than the 155 participants enrolled in the study since this was a dose-escalation study and adverse events occurred at all dose levels.
Arm/Group | Octreotide 40 mg | Octreotide 60 mg | Octreotide 80 mg
All-Cause Mortality (participants affected / at risk) | 1/155 | 0/91 | 1/58
Serious Adverse Events (participants affected / at risk) | 9/155 | 7/91 | 8/58
Other Adverse Events (participants affected / at risk) | 103/155 | 51/91 | 31/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Octreotide 40 mg (N=155) | Octreotide 60 mg (N=91) | Octreotide 80 mg (N=58)
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Transient ischemic attack (Nervous system disorders) | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0
Corneal abscess (Infections and infestations) | 1 | 0 | 0
Herpes simplex ophthalmic (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Intervertebral disc protusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Impaired healing (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Spleen disorder (Blood and lymphatic system disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Octreotide 40 mg (N=155) | Octreotide 60 mg (N=91) | Octreotide 80 mg (N=58)
Abdominal distension (Gastrointestinal disorders) | 7 | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 7 | 1
Abdominal pain upper (Gastrointestinal disorders) | 10 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 18 | 11 | 4
Dyspepsia (Gastrointestinal disorders) | 11 | 2 | 1
Flatulence (Gastrointestinal disorders) | 10 | 1 | 2
Nausea (Gastrointestinal disorders) | 30 | 14 | 6
Vomiting (Gastrointestinal disorders) | 4 | 3 | 4
Asthenia (General disorders) | 27 | 11 | 8
Oedema peripheral (General disorders) | 19 | 8 | 5
Cholelithiasis (Hepatobiliary disorders) | 4 | 3 | 3
Influenza (Infections and infestations) | 6 | 4 | 3
Nasopharyngitis (Infections and infestations) | 5 | 4 | 5
Upper respiratory tract infection (Infections and infestations) | 6 | 2 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 | 20 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3
Dizziness (Nervous system disorders) | 8 | 1 | 2
Headache (Nervous system disorders) | 44 | 18 | 20
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 23 | 9 | 6
Hypertension (Vascular disorders) | 6 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study cannot be published for a period of up to 150 days, 60 days for sponsor review and 90 days for patent protection. In addition, the first publication may only occur after the first multi-center publication or, if no such multi-center publication is made, 12-18 months after completion of the study at all study sites.